CLINICAL TRIAL: NCT04393259
Title: The Tommy's National Rainbow Clinic Study: Evaluation of a Specialist Antenatal Service for Women and Families Following a Stillbirth or Neonatal Death
Brief Title: The Tommy's National Rainbow Clinic Study
Status: Recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Dr Alexander Heazell, Professor of Obstetrics, University of Manchester
Other Study IDs: IRAS249991
Record Dates: First submitted 2020-05-13; First posted 2020-05-19 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Stillbirth
Keywords: Pregnancy after loss; Antenatal care; Anxiety; Depression
MeSH Terms: conditions — Stillbirth; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants: Women attending an antenatal service using the Rainbow Clinic model of care.
  Interventions: Other: Rainbow Clinic Model of Antenatal Care

INTERVENTIONS:
Other: Rainbow Clinic Model of Antenatal Care — Rainbow Clinic Model is an antenatal model of care with initial ultrasound scan at 23 weeks' gestation including uterine artery Doppler, frequency of subsequent scans determined using data from this initial scan. Continuity of care is provided by obstetricians and midwives.

SUMMARY:
The death of a baby before or shortly after birth affects approximately 1 in every 250 pregnancies in the UK meaning that over 4,000 parents experience the death of a baby each year in the UK. The majority of women who have experienced the loss of a baby will have another pregnancy, usually within a year.

Our analysis of 14 studies concluded that parents need specialist support from doctors and midwives in a future pregnancy to reduce the risk of pregnancy complications and to provide the care and support they need. The Rainbow Clinic model aims to provide specialist care and support to families who have experienced the death of a baby during pregnancy or shortly afterwards. Rainbow Clinic was initially established in St Mary's Hospital, Manchester in 2013.

The Rainbow Clinic team are now working to establish Rainbow Clinics in other maternity units throughout the UK. As this is a new clinical service the investigators would like to evaluate the care provided in the Rainbow clinics across the United Kingdom, to look at women's experiences of care, their levels of anxiety and depression, to identify where care can be improved and the pregnancy outcomes of women attending Rainbow Clinic. This evaluation needs information about pregnancy outcomes and women's experiences. Participation in this research study will allow us to collect and aggregate this information. The investigators will ask all women attending participating Rainbow Clinics to complete a short questionnaire early in their pregnancy and again at the end. The study will collect information about the outcome of their pregnancy.

DETAILED DESCRIPTION:
In the UK, 1 in 300 parents will experience a stillbirth each year, which is over 2,700 babies per year (Manktelow, Smith et al. 2016). There are also over 1,250 neonatal deaths per year, meaning there are approximately 4,000 bereaved families per year in the UK. The death of a baby before or shortly after birth is a profoundly distressing experience for women and their families and is invariably followed by a period of protracted grief (Heazell, Siassakos et al. 2016). Previous stillbirth or neonatal death is consistently recognised to increase parents' anxiety, emotional vulnerability and decrease confidence in the next pregnancy (Mills, Ricklesford et al. 2014). This is a cause for concern because studies in the general maternity population have suggested that elevated maternal anxiety increases the risk of adverse pregnancy outcomes, notably preterm birth and low birthweight (Black, Shetty et al. 2008). A recent UK longitudinal study reported that the negative psychological impacts of perinatal loss persist far beyond the next pregnancy and despite the birth of a healthy child (Blackmore et al., 2011). This may have significant long term effects on outcomes for subsequent children; previous history of stillbirth or neonatal death has been reported to disrupt maternal attachment and negatively impact on parenting (Warland, O'Leary et al. 2011). Many parents feel robbed of the 'normal' positive feelings they expected and have described to us how their subsequent pregnancies were characterised by heightened anxiety and fear (Mills, Ricklesford et al. 2014). Common misconceptions, such as the belief that a new pregnancy helps to 'get over' grief for a lost child, effectively isolates parents from social support networks, increasing reliance on external and professional intervention.

Qualitative studies of women's experiences of subsequent pregnancies highlight the value placed on regular interaction with health professionals (Côté-Arsenault, Donato et al. 2006, Côté-Arsenault 2007, Cote-Arsenault and Donato 2011). This evidence suggests that specialist antenatal support might ameliorate anxiety, improve experiences of pregnancy, support relationships and positively impact on future parenthood (Caelli, Downie et al. 2002). However, there is a dearth of evidence regarding what additional antenatal support parents' desire following a previous stillbirth or neonatal death.

To address the need for increased antenatal surveillance and support the Rainbow Clinic was established in St Mary's Hospital, Manchester in 2013 and rolled out in a neighbouring hospital in Manchester in 2016. An extensive quality improvement project and accompanying research study demonstrated that attendance at the Rainbow clinic improved pregnancy outcomes, decreased anxiety levels and was associated with a social value of £6.10 for each £1 invested. The investigators are now working to establish Rainbow Clinics in other maternity units. As this is a new clinical service there is a need to evaluate the care provided in the Rainbow clinics across the United Kingdom, to look at women's experiences of care, where care can be improved and its impact upon pregnancy outcomes for mothers and babies. This needs information about pregnancy outcomes and women's experiences. Participation in this research study will allow us to collect and aggregate this information.

ELIGIBILITY:
Inclusion Criteria:

* Women who are attending the Rainbow Clinic because they have had prior stillbirth, neonatal death or late termination of pregnancy
* Women who are currently pregnant

Exclusion Criteria:

* Less than 16 years of age
* Anyone who lacks capacity to consent

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pregnant women once booked for antenatal care, will be eligible for the study if they are attending the Rainbow clinic or equivalent service at one of the recruiting sites across the country.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Gestation of birth | At birth
  Gestation at birth in present pregnancy
Mode of birth | At birth
  Mode of delivery in present pregnancy
Admission to Neonatal Unit | At birth
  Admission to neonatal unit following delivery of the baby
Birthweight | At birth
  Recorded weight at birth

SECONDARY OUTCOMES:
Maternal Anxiety | 17 and 36 weeks' gestation
  Anxiety as assessed by Generalised Anxiety Disorder (2-item) (Lowest score 0 and Highest score 6, Higher score = more anxiety) and Cambridge Worry Score (Lowest score 0 and Highest score 85, Higher score = more worry).
Maternal Depression | 17 and 36 weeks' gestation
  Depression as assessed by Edinburgh Postnatal Depression Score (Lowest score 0 and Highest Score 30, Higher score = greater depression).

OTHER OUTCOMES:
Women's experience of care | 36 weeks' gestation
  Measured by bespoke patient experience questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No IPD plan

REFERENCES:
- [Derived] Barron RL, Tomlinson E, Bailey E, Heazell AE. Tommy's National Rainbow Clinic Study: a protocol for a multi-site cohort study to evaluate a specialist antenatal service for women and families following a stillbirth or neonatal death. BMJ Open. 2025 Aug 5;15(8):e103294. doi: 10.1136/bmjopen-2025-103294. PMID 40764070